CLINICAL TRIAL: NCT05943405
Title: The Disease Severity In Patients With Psoriasis
Status: Completed | Type: Observational
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Nurhasan Agung Prabowo, MD, Head of Hospital Research Unit, Universitas Sebelas Maret
Other Study IDs: NAP07
Record Dates: First submitted 2023-06-25; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Psoriasis
Keywords: Psoriasis; Psoriasis Area and Severity Index; Gamma-Glutamyl Transferase; CRP; Apolipoprotein B
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — 5 cc of blood was drawn for GGT, hs-CRP, and apo B examinations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to evaluate new markers to predict disease activity in psoriasis. The main question is SGOT, SGPT, GGT, hs-CRP, and apo B related to disease severity in psoriasis.

DETAILED DESCRIPTION:
Psoriasis patients who had signed an informed consent were assessed for PASI scores and 5 cc of blood was drawn for GGT, hs-CRP, and apo B examinations. A PASI score is a tool used to measure the severity and extent of psoriasis. PASI is an acronym for Psoriasis Area and Severity Index.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Psoriasis

Exclusion Criteria:

* Heart Failure
* Diabetes Mellitus
* Kidney Disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Psoriasis Patients
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Gamma-Glutamyl Transferase | only in admission
  Gamma-Glutamyl Transferase was check in admission, reference range for adults is 5 to 40 U/L (units per liter)
Apolipoprotein B | only in admission
  Apolipoprotein B (ApoB) is the primary apolipoprotein and is the carrier for the following lipids: chylomicrons, low-density lipoprotein ( LDL), very low-density lipoprotein (VLDL), intermediate-density lipoprotein (IDL), and lipoprotein. Unit used in mg/dL
High-sensitivity c-reactive protein | only in admission
  High-sensitivity C-reactive protein (hsCRP) is a marker of inflammation that predicts incident myocardial infarction, stroke, peripheral arterial disease, and sudden cardiac death. Unit used in mg/L
PASI | only in admission
  A PASI (The Psoriasis Area and Severity Index) score can range from 0 to 72

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Sebelas Maret Hospital, Sukoharjo, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sholihah MM, Kusuma TRH, Hanif MI, Prabowo NA. Letter to the Editor on Type 1 diabetes onset triggered by COVID-19. Acta Diabetol. 2021 Sep;58(9):1283-1284. doi: 10.1007/s00592-021-01761-3. Epub 2021 Jun 28. No abstract available. PMID 34181079
- [Result] Pratama YS, Pradiptakirana R, Rachmah A, Prabowo NA. Autoimmune Thrombocytopenia in SLE and COVID-19. Eur J Case Rep Intern Med. 2021 Nov 3;8(11):002863. doi: 10.12890/2021_002863. eCollection 2021. PMID 34912736